CLINICAL TRIAL: NCT07142681
Title: Changes in the Dietary Patterns of Adults in Family Units With a Newly Diagnosed Type 1 Diabetes Mellitus Child: Impact of Educational Actions Derived From Standard Care
Brief Title: Changes in the Dietary Patterns of Adults in Care of a Newly Diagnosed Type 1 Diabetes Mellitus Child
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital Sant Joan de Deu (Other); Hospital Arnau de Vilanova (Other); Fundació Institut de Recerca del Hospital Santa Creu i Sant Pau (Unknown)
Responsible Party: Principal Investigator, Joana Rossell, postdoctoral researcher, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: IIBSP-DDM-2023-166
Record Dates: First submitted 2025-07-02; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Dietary Habits; Parents; Diabetes Mellitus, Type 1
Keywords: diet; dietary habits; nutritional intervention; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Feeding Behavior; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to compare the feeding pattern evolution in parents whose children have been newly diagnosed with type 1 diabetes mellitus, versus one year later. The main question it aims to answer is:

- Does the dietary intervention in the pediatric population affect the parent's diet?

DETAILED DESCRIPTION:
Parents with newly diagnosed type 1 diabetes infant will be identified upon hospital admission.

Parents will be informed about the study and asked if they are willing to participate. If affirmative, the participant parent will sign the informed consent, and one of the investigators will hand over the different questionnaires. A brief physical exploration will be performed.

After one year, and coinciding with any programmed visit to the hospital, questionnaires will be handed over again, together with the repetition of the brief physical exploration.

The questonnairs include: Food register, Mediterranean adherence, physical activity, pediatric anxiety, and hospital anxiety and depression scale questionnaires.

Data will be extracted from the questionnaires, and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Parents or legal tutors of a child with type 1 diabetes (according to ADA criteria).
* Less than 1 week since the type 1 diabetes diagnostic.
* Living together more than 40%of the time with the infant with type 1 diabetes.
* Be the adult responsible for most of the family meals.

Exclusion Criteria:

* Parents of infants with other types of diabetes (type 2, MODY, gestational, others).
* Household members with diseases or conditions that can affect dietary habits (type 2 diabetes, kidney disease, pregnancies).
* Significant dietary habit modifications (change to a vegeterian, vegan, palea, or other diets, fasting situations) in the last month prior to the diagnosis of type 1 diabetes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parents of infants with recently diagnosed type 1 diabetes mellitus, that live most of the time with the infant, and are responsible for the household meals.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Food frequency estimation | 1 year
  Food and beverage consumption are evaluated with the deliverance of a Food Frequency Questionnaire tool - the Cuestionario de Frecuencia de Consumo de Alimentos (CFCA) - with 137 items and validated for the spanish population. A copy of the CFCA in english is attached in the protocol. Changes in portions, food items, and frequency can be estimated through the comparison of the questionnaire at basal and half time. The questionnaire evaluated will be the ones handled at the start and at the end of the study (0 and 12 months).
Adherence to Mediterranean Diet (Predimed questionnaire) | 1 year
  Predimed questionnaire, with 14 items and a punctuation associated to each answer answer, allowes the obtantion of a score. Obtaining a score of less than 9 indicates a poor adherence to the mediterranean diet, and obtaining a score of 9 or more indicates a good adherence to the mediterranean diet. English version: http://www.predimed.es/uploads/8/0/5/1/8051451/p14_meddiet_english_version.png The questionnaire evaluated will be the ones handled at the start and at the end of the study (0 and 12 months).

SECONDARY OUTCOMES:
Food frequency estimation (half time) | 6 months
  Food and beverage consumption are evaluated with the deliverance of a Food Frequency Questionnaire -the Cuestionario de Frecuencia de Consumo de Alimentos- (CFCA) with 137 items and validated for the spanish population. A copy of the CFCA in english is attached in the protocol.
  Changes in portions, food items, and frequency can be estimated through the comparison of the questionnaire at basal and half time.
  The questionnaire evaluated will be the ones handled at the start and half-time of the study (0 and 6 months).
Adherence to Mediterranean Diet (predimed) (half time) | 6 months
  Predimed questionnaire, with 14 items and a punctuation associated to each answer answer, allowes the obtantion of a score. Obtaining a score of less than 9 indicates a poor adherence to the mediterranean diet, and obtaining a score of 9 or more indicates a good adherence to the mediterranean diet. English version: http://www.predimed.es/uploads/8/0/5/1/8051451/p14_meddiet_english_version.png The questionnaire evaluated will be the ones handled at the start and half-time of the study (0 and 6 months).
Physical activity characterization | 6 and 12 months
  Evaluate the changes in the physyical activity during the first 6 months and the first year.
  Physical activity will be measured through the administration of the International Physical Activity Questionnaire (IPAQ). This questionnnaire contains 7 answers that gather information of vigourous and moderate activity, as well as walking. Each activity is multiplied by a standard unit for measuring energy expenditure (MET) which gives us information whether the physical activity of the subject is High, Moderate, or Low.
  The questionnaire will be handled at the start, half-time, and end of the study (0, 6, and 12 months).
Emotional stress characterization | 6 and 12 months
  Evaluate the changes in the emotional stress felt by the parents during the first 6 months and the first year.
  This outcome will be measured through the administration of the Hospital Anxiety and Depression Scale (HADS), consisting of 14 items, 7 for anxiety measurement and 7 for depression measurement. Each item can score between 0 to 4 points, with a maximum score for each subscale: 21. The two subscales score independently: 0-7 is normal, 8-10 borderline abnormal (mild), and over 11 abnormal (clinical case).
  The questionnaire will be handled at the start, half-time, and end of the study (0, 6, and 12 months).
Emotional impact of the diagnosis characterization | 6 and 12 months
  Evaluate the changes in anxiety and depression scale levels during the first 6 months and the first year.
  This outcome is measured through the administration of the validated Pediatric Inventory for Parents (PIP), used to measure parental stress related to caring for a child with a chronic illness. It evaluates both the frequency and the difficulty of stressors that parents experience through 42 items analyzing the frequency and the difficulty of an item. Each item can obtain a score between 0-5, and the final punctuation can range from 42 to 210, with higher punctuations indicating higher stress.
  The questionnaire will be handled at the start, half-time, and end of the study (0, 6, and 12 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

DOCUMENTS (1):
  • Study Protocol (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT07142681/Prot_000.pdf